CLINICAL TRIAL: NCT04568070
Title: Turkish Version of the Mini-BESTest: Transcultural Adaptation and Validation Study in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, Principal Investigator, Istanbul Medeniyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IMU Stroke
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Stroke; Balance; Distorted
Keywords: balance; stroke; validity; reliability
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke (Experimental): Stroke patients who applied to the Physical Medicine and Rehabilitation outpatient clinic, met the inclusion criteria and volunteered to participate in the study
  Interventions: Diagnostic Test: mini-BESTest (Mini-Balance Evaluation Systems Test); Diagnostic Test: Berg Balance Scale; Diagnostic Test: Timed Up and Go Test; Diagnostic Test: Functional Reach Test

INTERVENTIONS:
Diagnostic Test: mini-BESTest (Mini-Balance Evaluation Systems Test) — Balance evaluation test that has 14 tasks leading to a total possible score of 28 points requires only 10 to 15 minutes to conduct.
Diagnostic Test: Berg Balance Scale — The scale is a 14-item objective measure designed to assess static balance and fall risk in adult populations.
Diagnostic Test: Timed Up and Go Test — It is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Diagnostic Test: Functional Reach Test — The Functional Reach Test is a single item test developed as a quick screen for balance problems in older adults. A score of 6 or less indicates a significant increased risk for falls. A score between 6-10 inches indicates a moderate risk for falls.

SUMMARY:
"mini-BESTest (Turkish version)", "Berg Balance Test", "Timed Up and Go Test" and "Functional Reach Test" will be used for balance measurement in patients and the correlation of the mini-BEST with these tests will be checked.

DETAILED DESCRIPTION:
The first part of the study is the Turkish translation of mini-BESTest. After the translation process, "mini-BESTest (Turkish version)", "Berg Balance Test", "Timed Up and Go Test" and "Functional Reach Test" will be used for balance measurement in patients and the correlation of the mini-BEST with these tests will be checked. All tests will be applied by 2 researchers on the same day, 2 times with 10 minutes intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic stroke patients
2. Patients who can execute commands
3. Patients who are ambulatory enough to complete most balance tasks
4. Patients participating in the study voluntarily

Exclusion Criteria:

1. Acute stroke patients
2. Patients who cannot execute commands
3. Non-ambulatory patients
4. Pediatric patients and pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2020-12-24 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
mini-BESTest | 3 months
  Balance evaluation test that has 14 tasks leading to a total possible score of 28 points.
Berg Balance Scale | 3 months
  The scale is a 14-item objective measure designed to assess static balance and fall risk in adult populations
Timed Up and Go Test | 3 months
  It is a test used to assess a person's mobility and requires both static and dynamic balance
Functional Reach Test | 3 months
  The Functional Reach Test is a single item test developed as a quick screen for balance problems in older adults

CONTACTS AND LOCATIONS:
Overall Officials: Bilinç Karatekin, Principal Investigator — Istanbul Medeniyet University Physical Therapy And Rehabilitation Department
Locations (1):
- Istanbul Medeniyet University Faculty of Medicine, Physical Medicine and Rehabilitation Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No